CLINICAL TRIAL: NCT00253877
Title: A Prospective, Multi-Centre, Historical Control Trial Comparing the Conserve® Plus Resurfacing Hip System to Standard Total Hip Arthroplasty.
Brief Title: A Comparison of a Resurfacing Hip System to Standard Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OHREB 2003137-01H
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Hip Resurfacing
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conserve Plus Hip Resurfacing (Active Comparator): Conserve Plus Hip Resurfacing group. Complication rate will be compared between groups.
  Interventions: Other: Complication rate
- Total Hip Replacement (Other): Historical Total Hip Replacement control group of recently published conventional total hip replacement results (Williams, 2002). Complication rate will be compared between groups.
  Interventions: Other: Complication rate

INTERVENTIONS:
Other: Complication rate — All patients in the active comparator group received the Conserve Plus Hip Resurfacing System, manufactured by Wright Medical Technology. The complication rate and clinical efficacy will be recorded and compared to the Total Hip Replacement historical control group.

SUMMARY:
This study compares outcomes and metal ion levels between patients who receive the Conserve® Plus Hip System compared to those who have received a standard hip replacement in a recent study.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is currently the standard of care for end-stage degenerative joint disease of the hip. In this surgery, the entire joint is replaced by inserting an acetabular component into the pelvis, a femoral stem down the thigh bone (which has a ball on it to articulate in the acetabulum). However for the younger patient, long-term fixation and the prospect of multiple revisions remain a notable concern. Long-term results of THA in this patient population have been disappointing. Studies cite failure rates of 21% to 33% at less than 10 years follow up. The Conserve Plus Hip System differs from total hip arthroplasty as it uses less bone stock from the femoral bone. The prosthesis is designed so that the head of the femoral bone is resurfaced rather than replaced. Consequently, bone stock of the femur is conserved. The bone conserving nature of this implant allows the surgeon to convert to a total hip arthroplasty with ease should a time arise when the patient requires revision arthroplasty. The Conserve Plus Hip System is also different from the THA as the bearing surface is metal on metal, rather than the conventional metal on polyethylene. This metal on metal bearing surface provides lower wear. Theoretically, this type of hip replacement may be a viable alternative to THA for the younger patient.

ELIGIBILITY:
Inclusion Criteria:

- Patients who are undergoing primary hip surgery for noninflammatory degenerative joint disease (NIDJD). Composite diagnoses for NIDJD include osteo/degenerative arthritis, traumatic arthritis, congenital hip dysplasia, and avascular necrosis.2. Patients who are skeletally mature or at least 18 years of age.3. Patients for whom there is a reasonable expectation that they will be available for each examination scheduled over a two year post-operative follow up period and for annual exams until the last patient entered into the study has achieved two years of follow-up.4. Patients who agree to participate and sign the informed consent form.5. Patients who do not meet any of the exclusion criteria.6. Patients who are already enrolled in the study and present with a need for revision of the metal femoral or acetabular resurfacing components. These patients may have the failed component(s) revised with an investigational component.

Exclusion Criteria:

* . Patients who are less than 18 years of age or are skeletally immature at the time of surgery.2. Patients who present with inflammatory degenerative joint disease or revision surgery other than that specified in the inclusion criteria.3. Patients with previous fusions, acute femoral neck fractures and above knee amputations.4. Patients with evidence of active infection.5. Patients who are pregnant (or plan on becoming pregnant) or who are lactating.6. Patients with neurologic or musculoskeletal disease that may adversely affect gait or weight bearing.7. Patients who have previously undergone an ipsilateral hemi resurfacing, total resurfacing, total bipolar, unipolar, or total hip replacement device.8. Patients with active hepatitis or HIV infection.9. Patients who otherwise meet the study criteria, but refuse to consent in writing to participate in the study. 10. Patients who are obese where obesity is defined as a Body Mass Index (BMI) >35.11. Patients with neuropathic joints.12. Patients with severe documented psychiatric disease.13. Patients requiring structural bone grafts.14. Patients with a documented allergy to cobalt chromium molybdenum.15. Patients with ipsilateral girdlestone.16. Patients with sickle cell disease.17. Patients with significant femoral head or neck deformity or significant acetabular wall deficiency.18. Patients with renal impairment where renal impairment is defined as serum creatinine> 180umol/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-07 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Rate of complications | 2 years
  Any complications pertaining specifically to the implant

SECONDARY OUTCOMES:
Survivorship rate Clinical efficacy (Pain, Function, Radiographic outcome and Patient Satisfaction) Blood and Urine Ion Levels | 2 years
  Clincial efficiency pertaining to the implant directly

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kim, MD, FRCS(C), Principal Investigator — OHRI
Locations (3):
- Canada (3):
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec

REFERENCES:
- [Result] Kim PR, Beaule PE, Laflamme GY, Dunbar M. Causes of early failure in a multicenter clinical trial of hip resurfacing. J Arthroplasty. 2008 Sep;23(6 Suppl 1):44-9. doi: 10.1016/j.arth.2008.05.022. PMID 18722302